CLINICAL TRIAL: NCT05135832
Title: Patient Reported Outcomes by Patients With Metastatic Renal Cell Carcinoma; a Randomized Controlled Trial
Brief Title: Patient Reported Outcomes by Patients With Metastatic Renal Cell Carcinoma
Acronym: PRORECECA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Ida Rasmussen, Principal investigator, MD, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UR 2134; P-2021-693 (Other: Videnscenter for Dataanmeldelser / PACTIUS)
Record Dates: First submitted 2021-10-27; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Renal Cell Carcinoma; Kidney Cancer; Kidney Neoplasm; Urologic Cancer; Urologic Neoplasms; Advanced Renal Cell Carcinoma
Keywords: Patient-reported outcomes; Electronic reporting of symptoms; Physical function
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-reported outcomes arm (experimental arm) (Experimental): This arm will be assigned to intervention by weekly electronic reporting of symptoms and side effects in an app. A specifically developed alert-algorithm will in real-time guide the patient to adjust supportive care or contact the hospital.
  The reported symptoms are sent to the hospital to a healthcare professional - depending on the severity of the reported symptoms the healthcare professional can schedule a visit at the clinic.
  The patient will also receive a health-related quality of life questionnaire (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire) including the Physical Function domain in the app each month.
  Patient satisfaction regarding the patient-reported outcomes will be measured with the validated Patient-Reported Experience Measurement questionnaire at termination of participation.
  Interventions: Device: Electronic patient-reported outcomes regarding symptoms and health-related quality of life
- Standard of care (No Intervention): This arm will continue standard procedure regarding side effect registration and handling.
  The patients will receive a health-related quality of life questionnaire (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire, EORTC QOL-C30) at baseline, after 1, 3, and 6 months of participation in the study.

INTERVENTIONS:
Device: Electronic patient-reported outcomes regarding symptoms and health-related quality of life — Weekly reporting of patient-reported outcomes for closer contact between patient and clinic between treatment cycles.
  The supportive care (including drugs) is similar in the two treatment arms except for the use of electronic patient-reported outcomes.
  Other Names: ePRO; Alert-algorithm; active patient-reported outcomes; Real-time guidance of patients when symptom reporting
  Arms: Patient-reported outcomes arm (experimental arm)

SUMMARY:
The purpose of PRORECECA is to test whether adding weekly active patient-reported outcomes to the treatment of patients with metastatic renal cell carcinoma can improve patient-reported physical function.

DETAILED DESCRIPTION:
PRORECECA is a two-armed randomized controlled trial for patients with metastatic renal cell carcinoma initiating 1st or 2nd line of standard therapy.

Patients will be randomized to either receiving questions from Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE™) with a specifically developed alert-algorithm and the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) or receiving standard procedure regarding side effect registration and handling.

The hypothesis is that weekly active patient-reported outcomes in the intervention group can improve physical function 30% compared to the group who receive standard care and standard handling of side effects.

A total of 174 patients will be included with 87 patients in each arm.

Primary endpoint is physical function reported by the patient after 3 months of treatment. The patients will assess their physical function by completing the EORTC QLQ-C30.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic renal cell carcinoma
2. Age ≥ 18 years
3. Starting 1st or 2nd line treatment at enrolment
4. Performance status (PS) ≤ 2
5. Able to read Danish
6. No serious cognitive impairment
7. Patient has given written informed consent

Exclusion Criteria:

1. No smart phone
2. Patient participating in other interventional studies. This is only relevant for studies that might interfere with the intervention. Cases of doubt will be settled by the protocol committee.
3. Persons deprived of liberty or under guardianship or curators
4. Dementia, mental alteration or psychiatric disease that can compromise informed consent from the patient and / or adherence to the protocol and the monitoring of the trial
5. Earlier participation in PRORECECA (e.g. when changing from 1st to 2nd line of treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2021-12-13 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Physical function | Within the first 3 months of treatment
  Patient-reported physical function in the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) - Whether patients using PRO experience a better physical function compared to patients receiving standard care and handling of side effects.

SECONDARY OUTCOMES:
Health related quality of life | Within the first 6 months of treatment
  Registration of differences in quality of life between the two arms in the study.
  The quality of life questionnaires EORTC QLQ-C30 (scale range 0-100, a higher score indicating better quality of life) will be used for as quality of life measurement.
  Differences between the two arms will be tested using t-test and analysis of covariance (ANCOVA).
Admissions (number) | Within the first 6 months of treatment
  Registration of number of admissions. The registration is made to investigate whether the use of PRO and thereby a closer contact to the clinic between visits can decrease the number of hospital admissions.
Admissions (length) | Within the first 6 months of treatment
  Registration of length of admissions. The registration is made to investigate whether the use of PRO and thereby a closer contact to the clinic between visits can decrease the length of hospital admissions.
Symptom management (number) | Within the first 6 months of treatment
  Registration of differences in number of intervention in the two treatment arms.
Symptom management (type) | Within the first 6 months of treatment
  Registration of differences in types of intervention in the two treatment arms.
Number of contacts to the clinic | Within the first 6 months of treatment
  Registration of number of contacts to the clinic (both phone and attendance). The registration is made to investigate whether the use of PRO de- or increases the number of contacts to the clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Ida Marie L Rasmussen, MD, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Department of Oncology, Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No